CLINICAL TRIAL: NCT06810557
Title: Feasibility and Preliminary Efficacy of a Brief Behavioral Sleep Intervention for Excessive Weight Gain Prevention in Primary Care
Brief Title: Brief Behavioral Sleep Intervention for Obesity Prevention in Primary Care
Acronym: Rx SLEEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01DK139665 (NIH); R01DK139665 (NIH)
Record Dates: First submitted 2025-01-21; First posted 2025-02-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Obesity, Childhood; Short Sleep; Obesity Prevention
Keywords: sleep; behavioral intervention; primary care; obesity prevention; child; pediatric
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Sleep Intervention (Experimental): Behavioral intervention to enhance school-aged children's sleep
  Interventions: Behavioral: Optimize Sleep Primary Care (OSPC)
- Sleep Education (Other): Sleep Education
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Optimize Sleep Primary Care (OSPC) — In addition to standard care within Temple University Primary Care (TUPC), two face-to-face zoom sessions and four brief phone follow-ups (two during active treatment and two during maintenance) that focus on using effective behavioral strategies (e.g., goal setting, self-monitoring, positive reinforcement, stimulus control, problem-solving) to enhance children's sleep by approximately one hour/night.
  Arms: Behavioral Sleep Intervention
Other: Enhanced Usual Care — In addition to standard care within Temple University Primary Care (TUPC), the provision of six education contacts regarding children's sleep needs and the benefits of getting a good night's sleep.
  Arms: Sleep Education

SUMMARY:
The goal of this study is to compare two different approaches to help families with children 6-11 years enhance nighttime sleep: 1) working one-on-one with a nurse to learn effective behavioral strategies to try to improve children's sleep or 2) receiving education on a good night's sleep and its benefits. Participating families will meet with a nurse 6 times or receive 6 educational handouts. Participating families will also complete three assessments (start of the study, 2 months and 6 months) during which study questionnaires will be completed, participating children will wear devices that assess sleep and physical activity, participating families will report on what the child ate on two separate days and will be measured for height and weight.

DETAILED DESCRIPTION:
The present study is assessing the feasibility and preliminary effectiveness of a brief behavioral intervention to enhance children's sleep and prevent development of obesity. Fifty short sleeping (< 9 hours/night) children 6-11 years old who are primarily AA/Black and from lower socioeconomic backgrounds will be enrolled into a 6-month study. Children will be randomly assigned to 1 of 2 conditions: 1) optimize sleep primary care (OSPC; behavioral intervention to enhance sleep duration delivered by a nurse in primary care) or 2) enhanced usual care (EUC; usual care plus sleep education). All children will receive standard pediatric care. Families randomized to OSPC will receive a four-session intervention (two zoom-delivered sessions and two brief phone follow-ups) over the first two months with two additional phone follow-ups during maintenance (months 2-6). Families randomized to EUC will receive sleep education that is delivered at the same points of contact as OSPC sessions. At baseline, end of treatment (2 months), and 6 months, the following will be measured from a Reach, Effectiveness, Adoption, Implementation, Maintenance (RE-AIM) perspective: reach (e.g., enrollment), adoption (e.g., pediatric provider engagement), implementation (e.g., session attendance, treatment fidelity), maintenance (e.g., retention), and preliminary effectiveness (e.g., changes in sleep duration (actigraphy), eating behaviors (24-hour dietary recalls), physical activity (accelerometry), and anthropometrics (measured height and weight).

ELIGIBILITY:
Inclusion Criteria:

* Patient at Temple Pediatrics
* Child age 6-11 years
* Child time in bed of less than 9 hours per night on most days per week
* Body Mass Index (BMI) for age and biological sex great than the 10th percentile but less than the 95th percentile
* Understanding of and ability to complete the protocol
* Parent age at least 18 years and primary caregiver
* Willingness to be randomized to either condition

Exclusion Criteria:

* Diagnosed sleep disorder
* Medication use or diagnosis of medical or psychiatric condition that may impact sleep or weight status
* Current or planned treatment for weight control

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Achievement of enrollment goal | baseline
  Primary variable of interest is achievement of a priori goals for study enrollment (i.e., whether 50 families enroll in the study). We will also explore: of children referred, the number who enroll; and of children who are referred and eligible, the number who enroll.
The number of providers who participate and refer to the intervention | baseline
  Of all pediatric providers in the clinic, the number who attend the initial in-service training and the number of referrals each provider makes to the program. Attendance and the number of referrals will be tracked by study staff.
Average family attendance at intervention sessions | baseline to 6 months
  Whether or not families attend each treatment sessions will be captured by the study nurse. Primary variable of interest is whether families, on average, achieve > 75% attendance at all intervention sessions.
Nurse percent fidelity/accuracy in delivering the intervention | baseline to 6 months
  All intervention sessions are recorded to determine the accuracy with which nurses deliver the intervention. Specifically, trained staff review recordings and use a checklist to mark whether or not each intervention component is delivered during each session. Primary variable of interest is whether the nurse delivers the intervention with at least 80% fidelity/accuracy.
Percent of families who are retained in the study at both follow-up time points | baseline to 6 months
  Retention at both 2- and 6-months will be tracked by study staff and compared across study arms with a goal of at least 80% retention at two months.
Family assessment of the intervention's acceptability | baseline to 6 months
  Acceptability will be measured by families' responses to the overall acceptability question on the Theoretical Framework for Acceptability (TFA) Acceptability Scale. Specifically, families use a 5-point, likert-type scale ranging from 'completely unacceptable' to 'completely acceptable' to rate the intervention. The percent of families who rate the intervention as 'acceptable' or 'completely acceptable' will be assessed with a goal of at least 80% of families rating it as such.

SECONDARY OUTCOMES:
Preliminary Effectiveness: Sleep | baseline to 6 months
  Measured with actigraphy over 7 days at each assessment and scored with the assistance of sleep diaries and call-ins to time-stamped voicemail. Primary variable of interest is change in the actigraph-estimated sleep period, which is the time between actigraph-estimated bedtime and wake time.
Preliminary Effectiveness: Weight Status | baseline to 6 months
  Child height and weight will be measured by staff to calculate body mass index (BMI). Change in BMI (controlling for child age and biological sex) is of primary interest.
Preliminary Effectiveness: Diet - Caloric Intake | baseline to 6 months
  Measured with 24-hour dietary recalls on two days (one weekday and one weekend day). Mean reported caloric intake will be computed.
Preliminary Effectiveness: Diet - Percent Calories from Fat | baseline to 6 months
  Measured with 24-hour dietary recalls on two days (one weekday and one weekend day). Mean reported percent calories from fat will be computed.
Preliminary Effectiveness: Physical Activity | baseline to 6 months
  Measured with hip-worn accelerometry. Time spent in moderate to vigorous physical activity (controlling for wear time) is of primary interest.
Preliminary Effectiveness: Sedentary Activity | baseline to 6 months
  Measured by parent and child report during 24-hour dietary recalls (one weekday and one weekend day). Mean hours of TV viewing is of primary interest.

CONTACTS AND LOCATIONS:
Overall Officials: Chantelle N Hart, PhD, Principal Investigator — Temple University
Locations (1):
- Temple Pediatrics, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified, cleaned and scored summary data of the following will be shared: parent-completed surveys, child-worn actigraph and accelerometry data, staff-measured parent and child height and weight data, and staff-tracked process data
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available by the end of the award and will remain available for at least 5 years.